CLINICAL TRIAL: NCT05536076
Title: Effect of Hypercapnia Treatment on Respiratory Recovery After Spinal Cord Injury
Acronym: RECOV2SCI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: VA Detroit Healthcare System (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B4114-P
Record Dates: First submitted 2022-07-28; First posted 2022-09-10 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Sleep Apnea; SCI/D; Hypercapnia
Keywords: Sleep apnea; SCI/D; Hypercapnia
MeSH Terms: conditions — Sleep Apnea Syndromes; Hypercapnia

STUDY DESIGN:
Intervention Model Description: Controlled pilot trial to assess the feasibility of using daily chemical stimuli (acute intermittent hypercapnia) in patients with chronic SCI/D in comparison to able-bodied patients with OSA.
Who Masked: Participant
Masking Description: Participants (SCI N=10, SD N=10 and Able bodied N=10) will be undergo the intervention arm (acute intermittent hypercapnia)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intervention hypercapnia arm (Active Comparator): Intermittent hypercapnia treatment five days per week for two weeks.
  Interventions: Other: Hypercapnia treatment
- SCD (Experimental): Intermittent hypercapnia treatment five days per week for two weeks.
  Interventions: Other: Hypercapnia treatment
- Able-Bodoed (Experimental): Intermittent hypercapnia treatment five days per week for two weeks.
  Interventions: Other: Hypercapnia treatment

INTERVENTIONS:
Other: Hypercapnia treatment — Intermittent hypercapnia treatment five days per week for two weeks.

SUMMARY:
It is estimated that 1,275,000 people in the United States alone live with spinal cord injury, including around 100,000 Veterans with spinal cord injury, making the V.A. the largest integrated health care system in the world for spinal cord injuries injury care. New therapies are needed to prevent the morbidities and mortalities associated with the high prevalence of respiratory disorders in Veterans with spinal cord injury. The current research project and future studies would set the base for developing innovative therapies for this disorder. This proposal addresses a new therapeutic intervention for sleep apnea in spinal cord injury. The investigators hypothesized that daily hypercapnia treatments improve respiratory symptoms and alleviate sleep apnea in patients with chronic spinal cord injury. The investigators will perform a pilot study to examine the impact of daily hypercapnia treatments for-two week durations among Veterans with spinal cord injury. The investigators believe that this novel approach to treating sleep apnea and will yield significant new knowledge that improves the health and quality of life of these patients.

DETAILED DESCRIPTION:
One of the most devastating consequences of cervical spinal cord injury (SCI) is damage to the phrenic motor network, controlling the diaphragm (primary muscle of breathing). Subsequent diaphragm paralysis or paresis results in life-threatening impairments in breathing and can necessitate a need for ventilator assistance. Respiratory and cardiovascular complications are the most common causes of death in the first year post-injury (51% combined). Thus, there is an urgent need to develop strategies for improving function for people with acute and chronic spinal cord injury. Currently, treatments for respiratory dysfunction in spinal cord injury patients are limited to mechanical devices or nerve pacing. Moreover, the proposed plan of studying respiratory muscle training in spinal cord injury patients is novel. However, it is based on animal and human studies that have shown with validity that respiratory muscle training using mild intermittent hypoxia improves respiratory function following SCI. However, the effect of intermittent hypoxia has shown to be dependent on the level of alveolar CO2 and may pose undesirable cardiovascular effects. Previous studies showed that respiratory recovery following SCI manifests by a delayed and partial restorative spontaneous plasticity. The current research project and future anticipated studies would set the base for developing innovative therapies that can stimulate respiratory plasticity hence recovery for this prevalent disorder.

The proposed pilot/feasibility study will test the effect of daily acute intermittent hypercapnia (dAIHc) in individuals with SCI. The objectives of this study are to (1) determine recruitment rates and test the feasibility of recruitment, (2) calculate withdrawal and dropout rates, (3) test the feasibility and tolerability and acceptability of the proposed intervention in an SCI population, (4) develop and refine a new respiratory training intervention using dAIHc paradigm (5) derive effect size estimates for clinical endpoints and their associated variability at the end of treatment to calculate an appropriate sample size for an adequately powered clinical trial. Compared to sham therapy, the central hypothesis is that the daily respiratory muscle training (dAIHc) approach is acceptable and feasible in patients with SCI and will strengthen respiratory muscles and reduce the severity of sleep-disordered breathing (SDB), and will improve daytime symptoms.

This study is highly innovative and the first of its kind in patients with SCI, as it seeks first to use a new set of rehabilitative exercises to improve ventilation and respiratory muscles strength; secondly, it aims to use controlled randomized design; finally, it will determine the role of respiratory muscle exercises in reducing the severity of sleep symptoms and daytime function in SCI. Each aim is independently testable and does not depend on the result of the other aims. The findings will likely apply to a broad range of other neuromuscular diseases (such as Multiple Sclerosis and Stroke). The team of this pilot project has the resources and IRB approval necessary to execute the project.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with chronic SCI/D (>6 months post-injury)
* American Spinal Injury Association (ASIA) classification A-D who have evidence of SDB (excluding those with no evidence of a neurologic deficit based on ASIA classification)
* Able-bodied patients (without SCI/D0 who have OSA.

Exclusion Criteria:

* Receiving continuous mechanical ventilation (except PAP therapy which is considered usual treatment for SDB
* Severe congestive heart failure with ejection fraction <35%
* Recent health event that may affect sleep
* stroke
* acute myocardial infarction
* recent surgery
* hospitalization
* Alcohol or substance abuse (<90 days sobriety)
* Self-described as too ill to engage in study procedures
* Evidence of hypercapnia on spontaneous breathing (end-tidal CO2 >50 mmHg)
* Unable to provide self-consent for participation

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | 2 weeks
  Determine the recruitment rate in the intervention arm and determine how many continue into the sham arm. (Number of patients enrolled and completed the study)

SECONDARY OUTCOMES:
Minute Ventilation | 2 weeks
  To measure the change in minute ventilation (L/min)
Change in sleep apnea severity | 2 weeks
  Severity of sleep apnea (Apnea-hypopnea index -events/hour)

CONTACTS AND LOCATIONS:
Overall Officials: Abdulghani Sankari, MD PhD, Principal Investigator — John D. Dingell VA Medical Center, Detroit, MI
Locations (1):
- John D. Dingell VA Medical Center, Detroit, MI, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
Publications from research will be made available to the public through the national Library of Medicine PubMed within one year after the date of publication. Final data sets underlying all publications resulting form the proposed research will be shared outside if the following criteria is met: A limited Dataset will be created and shared pursuant to Data Use Agreement (DUA) appropriately limiting use for dataset and prohibiting the recipient from identifying or re-identifying any individuals whose data are included in the dataset.
Supporting Information: Study Protocol, SAP
Time Frame: Within one year of the publication